CLINICAL TRIAL: NCT01117948
Title: A Multicentre Double-blind, Placebo-controlled, Randomised, Parallel-group Study to Evaluate the Efficacy and Safety of Lornoxicam in Patients With Mild to Moderate Probable Alzheimer´s Disease.
Brief Title: Efficacy and Safety of Lornoxicam in Patients With Mild to Moderate Probable Alzheimer´s Disease.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of Efficacy
Sponsor: JSW Lifesciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR081101/CO14950
Record Dates: First submitted 2010-05-04; First posted 2010-05-06 (Estimated); Results first posted 2012-11-29 (Estimated); Last update posted 2013-02-06 (Estimated); Status verified 2013-02

CONDITIONS: Alzheimer´s Disease
MeSH Terms: interventions — lornoxicam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lornoxicam (Experimental): Lornoxicam (8 mg) tablets to be taken orally two times daily (BID) for a period of 6 months.
  Interventions: Drug: Lornoxicam
- Placebo (Placebo Comparator): Placebo (8 mg) tablets to be taken orally two times daily (BID) for a period of 6 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lornoxicam — Lornoxicam (8 mg) tablets to be taken orally two times daily (BID) for a period of 6 months.
  Other Names: Xefo; Telos
  Arms: Lornoxicam
Drug: Placebo — Placebo (8 mg) tablets to be taken orally two times daily (BID) for a period of 6 months.
  Arms: Placebo

SUMMARY:
Study title: A multicentre double-blind, placebo-controlled, randomised, parallel-group study to evaluate the safety and efficacy of Lornoxicam in patients with mild to moderate probable Alzheimer's Disease.

Study phase: II

Indication: Alzheimer´s Disease

Investigational product, dose schedule and route of administration: Lornoxicam (8 mg) tablets to be taken orally two times daily (BID) for a period of 6 months.

Reference product, dose, schedule and route of administration: Placebo (8 mg) tablets to be taken orally two times daily (BID) for a period of 6 months.

DETAILED DESCRIPTION:
Study title: A multicentre double-blind, placebo-controlled, randomised, parallel-group study to evaluate the safety and efficacy of Lornoxicam in patients with mild to moderate probable Alzheimer's Disease.

Study phase: II

Indication: Alzheimer´s Disease

Study objectives: Primary:

To evaluate the efficacy of Lornoxicam (8 mg, BID) administered for 6 months versus matched placebo based on the following end-point:

• Cognitive performance - ADAS-cog+

Secondary:

To evaluate the efficacy of Lornoxicam (8 mg, BID) administered for 6 months versus matched placebo based on the following end-point:

* Activities of daily living - ADCS-ADL
* Behavioral / psychiatric symptoms - NPI

To evaluate the safety of Lornoxicam (8 mg, BID) administered for 6 months versus matched placebo.

• Overall incidence of adverse events.

Exploratory:

In a subgroup of 50 patients MRI analyses will be performed. In a subgroup of 50 patients exploratory data on the production of amyloid biological markers - blood plasma concentration of Aß1-38, Aß1-40 and Aß1-42 will be collected.

An optional 6 month open-label phase will be available.

Subject population, diagnosis and main criteria for inclusion: Male and female patients with mild to moderate probable Alzheimer's Disease according to NINCDS-ADRDA criteria

* Age 50 - 85 years inclusive
* MMSE 18-26 inclusive
* No history of treatment with Acetylcholine-esterase inhibitors or 4 weeks wash out period before baseline visit.
* No history of treatment with Memantine or 4 weeks wash out period before baseline visit.

Duration of treatment: 6 month double-blind phase 6 month open-label phase (optional)

Total number of subjects: A total of 220 patients will be recruited to the study from approximately 20 centers in a treatment ratio of 1:1 (8 mg BID, 110 : placebo, 110). This reflects the minimum number of patients required and also allows for a drop out rate of approximately 20%. Additional subjects may be recruited based on interim analysis.

Number of study centres: Approximately 20; multinational Europe

Number of visits: Doubble-Blind Phase: 5 visits (including screening); Open-Label Phase: 3 visits

Investigational product, dose schedule and route of administration: Lornoxicam (8 mg) tablets to be taken orally two times daily (BID) for a period of 6 months.

Reference product, dose, schedule and route of administration: Placebo (8 mg) tablets to be taken orally two times daily (BID) for a period of 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women (non-childbearing potential) with a diagnosis of Alzheimer's Disease according to the NINCDS-ADRDA clinical criteria.
2. Mild to moderate stage of Alzheimer's disease according to MMSE 18-26 inclusive.
3. Modified Hachinski Ischemic Scale equal to or below 4.
4. Geriatric Depression Scale below or equal 7.
5. If anticholinesterasic treatment had been prescribed, the patient must undergo a 4 week wash out period before the baseline visit (visit 1).
6. If Memantine treatment had been prescribed, the patient must undergo a 4 week wash out period before the baseline visit (visit 1).

Exclusion criteria:

1. Clinical, laboratory or neuroimaging findings consistent with:

* other primary degenerative dementia, (dementia with Lewy bodies, frontotemporal dementia, Huntington's disease, Jacob-Creutzfeld Disease, Down's syndrome, etc.)
* other neurodegenerative condition (Parkinson's Disease, amyotrophic lateral sclerosis, etc.)
* cerebrovascular Disease (major infarct, one strategic or multiple lacunar infarcts, extensive white matter lesions > one quarter of the total white matter)
* other central nervous system diseases (severe head trauma, tumors, subdural haematoma or other space occupying processes, etc.)
* seizure disorder
* other infectious, metabolic or systemic diseases affecting central nervous system (syphilis, present hypothyroidism, present vitamin B12 or folate deficiency confirmed by current analyses not older than 1 month, serum electrolytes out of normal range, juvenile onset diabetes mellitus, etc.) 2. A current DSM-IV diagnosis of active major depression, schizophrenia or bipolar disorder.

  3. Chronic daily drug intake for a time period of ≥ 14 days or expected for ≥ 14 days: "
* antidepressants, benzodiazepines, neuroleptics, major sedatives or other anti-inflammatory drugs including acetylic salicylic acid defined
* antiepileptics
* anticholinergics
* nootropics (including Ginkgo)
* centrally active anti-hypertensive drugs (clonidine, alpha-methyl dopa, guanidine, guanfacine,)
* opioid containing analgesics
* anti-inflammatory agents, cortico-steroids or immunosuppressants
* Cimetidin as gastroprotective drug 4. Severe thrombocytopenia defined as platelet counts <100.000 per mm3. 5. Coagulation disorders

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2009-09; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Sterner, M.Sc., Study Director — JSW-Life Sciences; Reinhold Schmidt, MD, Study Chair; Michael Rainer, MD, Principal Investigator

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient in: 09 Nov 2009 Last patient out: 30 Apr 2011 Patients were recruited in Clinics and Outpatient Clinics
Pre-assignment Details: Patients were excluded if they did not meet all inclusion/exclusion criteria or if the caregiver was not giving consent to participation in the trial
Period: Double Blind
Arm/Group | Lornoxicam | Placebo
Started | 111 | 108
Completed | 93 | 98
Not Completed | 18 | 10
Period: Open Label
Arm/Group | Lornoxicam | Placebo
Started | 93 | 98
Completed | 41 | 51
Not Completed | 52 | 47

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lornoxicam | Placebo | Total
Number analyzed (Participants) | 111 | 108 | 219
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 19 | 29
  >=65 years | 101 | 89 | 190
Age Continuous [Mean (Standard Deviation); unit: years] | 74.5 (6.75) | 73.6 (8.11) | 74.1 (7.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 67 | 136
  Male | 42 | 41 | 83
Region of Enrollment [Number; unit: participants]
  Austria | 35 | 35 | 70
  Czech Republic | 37 | 41 | 78
  Slovakia | 28 | 21 | 49
  Germany | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Cognitive Performance - ADAS-cog+
Description: Alzheimer's disease Assessment Scale, Cognitive Subscale (15 item) Higher scores indicate cognitive impairment. All items are assessed by independent rater (psychologists). The score goes from 0 points (no cognitive impairment) to 95 points (maximum impairment in all 15 items).
  Primary Outcome Measure is the change from baseline ADAS-cog+ score to the score after 26 weeks (end of double blind).
Time Frame: 6 months double blind, 6 months open-label (optional)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lornoxicam | Placebo
Number analyzed (Participants) | 93 | 98
units on a scale | -0.05 (6.75) | -0.89 (7.84)

2. Secondary Outcome: Activities of Daily Living - ADCS-ADL; Behavioral/Psychiatric Symptoms - NPI
Time Frame: 6 months double-blind, 6 months open label (optional)
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Lornoxicam | Placebo
Serious Adverse Events (participants affected / at risk) | 11/111 | 2/108
Other Adverse Events (participants affected / at risk) | 0/111 | 0/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lornoxicam (N=111) | Placebo (N=108)
Acute ulcus ventriculi (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal Ulcer with Bulb Stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
External abscess on the neck (Infections and infestations) | 0 (0) | 1 (1)
Gastric and duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Sudden death (General disorders) | 1 (1) | 0 (0)
Surgery of lumbar spine (Surgical and medical procedures) | 1 (1) | 0 (0)
Ulcus duodeni perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Syncope (Cardiac disorders) | 0 (0) | 1 (1)
Myocard infarction (Cardiac disorders) | 0 (0) | 1 (1)
Organic disorder with delusions (Psychiatric disorders) | 1 (1) | 0 (0)
Vertebral algic syndrom, Coxarthrosis - worsenig (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Local ischemy in right cerebellum hemisphera (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less